CLINICAL TRIAL: NCT01798511
Title: A Randomized Controlled Trial of Oral Refeeding Intolerance After Nasogastric Tube Feeding
Brief Title: Oral Refeeding IntOlerance After Nasogastric Tube Feeding (ORION)
Acronym: ORION
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Auckland, New Zealand (Other)
Responsible Party: Principal Investigator, Max Petrov, Principal Investigator Dr. Max Petrov, University of Auckland, New Zealand
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13/NTA/9
Record Dates: First submitted 2013-02-13; First posted 2013-02-26 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Acute Pancreatitis
Keywords: enteral nutrition; acute pancreatitis; oral food intolerance
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasogastric Tube Feeding (Experimental): Patients who are to have NTF will receive enteral nutrition within 6 hours after randomisation via a nasogastric tube placed into the stomach. A commercially available low fat semi-elemental feed (Peptisorb®, Nutricia Clinical NZ) will be used. The caloric target will be 2000 kcal per day. Enteral tube feeding will be commenced at a rate of 30 mL/h and increased gradually until 100 mL/h over 24-48 h.
  Interventions: Procedure: Nasogastric Tube Feeding
- Conventional Nutritional Management (Active Comparator): Patients who are to have CNM will be on nil-by-mouth regimen until they either develop signs of severe AP (in which case enteral tube feeding will be introduced) or the signs of AP mitigate,in which case clear liquids (as tolerated) followed by oral food (as tolerated) will be introduced.
  Interventions: Other: Conventional Nutritonal Management

INTERVENTIONS:
Procedure: Nasogastric Tube Feeding — A nasogastric tube will be placed into the stomach of patients.
  Arms: Nasogastric Tube Feeding
Other: Conventional Nutritonal Management — Patients who are to have CNM will be on nil-by-mouth regimen until they either develop signs of severe AP (in which case nasojejunal tube feeding will be introduced) or the signs of AP mitigate (in which case clear liquids (as tolerated) followed by oral food (as tolerated) will be introduced)
  Arms: Conventional Nutritional Management

SUMMARY:
Acute pancreatitis (AP) is one of the most common diseases in routine clinical practice of surgeons and gastroenterologists throughout the world. The high rate of pain relapse after oral refeeding contributes to high consumption of healthcare resources and prolonged hospital stay in AP patients. The data from the pilot MIMOSA trial suggest that early administration of nasogastric tube feeding may prevent pain relapse after oral refeeding in AP. The potential beneficial effects of enteral tube feeding include induction of postprandial gastrointestinal motility and improving the tolerance of oral refeeding. This may reduce the risk of pain relapse, thereby shortening length of hospital stay and reducing cost of treatment. The primary endpoint of the ORION trial will be the incidence of oral food intolerance. All eligible AP patients will be randomly allocated to either the Early Nasogastric Tube (ENT) group or Conventional Nutritional Management group (CNM) at 24h of hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AP
* Age 18 years or older
* Written informed consent
* Ongoing need for opiates

Exclusion Criteria:

* 96 hours after onset of symptoms
* Chronic pancreatitis
* Post-ERCP pancreatitis
* Intraoperative diagnosis
* Pregnancy
* Malignancy
* Received nutrition before randomisation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-04-01 (Estimated); Primary Completion 2015-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of oral food intolerance | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks

SECONDARY OUTCOMES:
Progression of severity | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Pain relapse | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Use of opioids | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks
Duration of hospital stay | Participants will be followed for the duration of hospital stay, an expected average of 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Max Petrov, MD, MPH, PhD, Principal Investigator — University of Auckland, New Zealand
Locations (1):
- University of Auckland, Auckland, New Zealand